CLINICAL TRIAL: NCT00772811
Title: Allogeneic Non-Myeloablative Stem Cell Transplantation Using Fludarabine and Melphalan Conditioning Regimen for Chronic Lymphocytic Leukemia, Lymphoma, and Multiple Myeloma
Brief Title: Using Fludarabine and Melphalan Conditioning Regimen for CLL,Lymphoma,Multiple Myeloma
Acronym: Flu-Mel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: Je-Hwan Lee, Asan Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-001
Record Dates: First submitted 2008-10-05; First posted 2008-10-15 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Lymphocytic Leukemia; Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flu-Mel (No Intervention): Conditioning chemotherapy before infusion of allogeneic stem cells will include fludarabine 30 mg/m2/day for 5 consecutive days (days -6 to -2) and melphalan 100 mg/m2 at day -2.
  Interventions: Drug: Flu-Mel

INTERVENTIONS:
Drug: Flu-Mel — * Fludarabine and Melphalan will be infused intravenously over 30 minutes in D5W 100 mL.
  * Melphalan will be administered following the completion of Fludarabine infusion at day -2.
  Other Names: Fludara-Alkaran

SUMMARY:
Allogeneic Non-Myeloablative Stem Cell Transplantation Using Fludarabine and Melphalan Conditioning Regimen for Chronic Lymphocytic Leukemia, Lymphoma, and Multiple Myeloma

DETAILED DESCRIPTION:
Treatment plan

* Conditioning chemotherapy before infusion of allogeneic stem cells will include fludarabine 30 mg/m2/day for 5 consecutive days (days -6 to -2) and melphalan 100 mg/m2 at day -2.
* Fludarabine and Melphalan will be infused intravenously over 30 minutes in D5W 100 mL.
* Melphalan will be administered following the completion of Fludarabine infusion at day -2.
* In case of unrelated donor HCT, thymoglobuline 3 mg/kg in N/S 500 mL (less than 0.5 mg/mL) or lymphoglobuline 15 mg/kg in N/S 500 mL (less than 2 mg/mL) IV qd on days -4, -3 and -2. Infuse over 4 hrs. Premedicate with Avil 45.5 mg IVP and Tylenol 600 mg po. Methylprednisolone 2 mg/kg in D5W 100 ml will be given IV over 30 minutes before thymoglobulin (or lymphoglobuline) on days -4 to -2.
* Before the administration of melphalan, prehydration will be done intravenously with 0.9% NS 1L over 3 hours.
* 30 minutes before melphalan infusion, premedication with dexamethasone 10 mg and ativan 1 mg i.v. push will be given. Appropriate antiemetics such as ondansetron 8 mg i.v. push every 4-6 hours and ativan 1-2 mg i.v. push every 4-6 hours will be administered.
* Hydration with 0.9% NS at 80 mL/hour will be administered for at least 7 days. Appropriate amount of KCl should be mixed.
* GVHD prophylaxis will include cyclosporine A (CSA) and methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 15 years of age or older and 65 years of age or younger
* Patients with CLL, lymphoma, or multiple myeloma will be included in this study
* No prior anti-cancer treatment should be done within 30 days.
* Informed consent should be given.
* Patients should have an HLA-identical or single HLA-locus mismatched donor.
* Karnofsky performance scale should be 50 or over (see Appendix I).

Exclusion Criteria:

* Patients must not have a psychiatric disorder or mental deficiency severe as to make compliance with the stem cell transplant treatment unlike, and making informed consent impossible.
* Patients with high serum creatinine level will be excluded.
* Patients should have uncontrolled infection.
* No major anticipated illness or organ failure incompatible with survival from stem cell transplant.
* Serum bilirubin less than or equal to 4.0 mg/dL.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2001-07; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate engraftment, chimerism, toxicity, incidence of acute graft-versus-host disease (GVHD), and day 100 treatment-related mortality (TRM) | 9years
  -To evaluate engraftment, chimerism, toxicity, incidence of acute graft-versus-host disease (GVHD), and day 100 treatment-related mortality (TRM) following allogeneic nonmyeloablative stem cell transplantation using fludarabine and melphalan conditioning regimen in patients with chronic lymphocytic leukemia (CLL), lymphoma, and multiple myeloma.

SECONDARY OUTCOMES:
include tumor response, incidence of chronic GVHD, and immune reconstitution. | 9years
  -The secondary objectives include tumor response, incidence of chronic GVHD, and immune reconstitution.

CONTACTS AND LOCATIONS:
Overall Officials: Je-Hwan Lee, Doctor, Principal Investigator — COSAH
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Lee JH, Kim DY, Seol M, Lee YS, Kang YA, Jeon M, Lee KH. A Phase II Trial of Fludarabine/Melphalan 100 Conditioning Therapy Followed by Allogeneic Hematopoietic Cell Transplantation for Patients With Lymphoma. Clin Lymphoma Myeloma Leuk. 2015 Nov;15(11):655-63. doi: 10.1016/j.clml.2015.08.087. Epub 2015 Sep 3. PMID 26428486
- See also: Flu-Mel — http://www.google.co.kr